CLINICAL TRIAL: NCT01879722
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Safety, Tolerability and Pharmacokinetic Study of Multiple Rising Doses of TAK- 063 in Subjects With Stable Schizophrenia and Healthy Japanese Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic Study of Multiple Rising Doses of TAK- 063 in Participants With Stable Schizophrenia and Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-063_104; U1111-1139-5355 (Other: World Health Organization)
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Results first posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Schizophrenia
Keywords: Drug therapy
MeSH Terms: conditions — Schizophrenia | interventions — 1-(2-fluoro-4-(1H-pyrazol-1-yl)phenyl)-5-methoxy-3-(1-phenyl-1H-pyrazol-5-yl)pyridazin-4(1H)-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- TAK-063 3 mg (Experimental): TAK-063 3 mg, tablets, orally, once daily for 7 days.
  Interventions: Drug: TAK-063
- TAK-063 10 mg (Experimental): TAK-063 10 mg, tablets, orally, once daily for 7 days.
  Interventions: Drug: TAK-063
- TAK-063 20 mg (Experimental): TAK-063 20 mg, tablets, orally, once daily for 7 days.
  Interventions: Drug: TAK-063
- TAK-063 30 mg (Experimental): TAK-063 30 mg, tablets, orally, once daily for 7 days.
  Interventions: Drug: TAK-063
- TAK-063 100 mg (Experimental): TAK-063 100 mg, tablets, orally, once daily for 7 days.
  Interventions: Drug: TAK-063
- Placebo (Placebo Comparator): Placebo matching TAK-063, tablets, orally, once daily for 7 days.
  Interventions: Drug: TAK-063 Placebo

INTERVENTIONS:
Drug: TAK-063 — TAK-063 tablets
  Arms: TAK-063 10 mg; TAK-063 100 mg; TAK-063 20 mg; TAK-063 3 mg; TAK-063 30 mg
Drug: TAK-063 Placebo — TAK-063 placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of TAK-063 when administered as multiple oral doses at escalating dose levels in participants with stable schizophrenia and in healthy Japanese participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-063. TAK-063 is being tested to find a well-tolerated dose and also to treat schizophrenia. This study will look at how well different doses of TAK-063 are tolerated in healthy people of Japanese descent and in people with stable schizophrenia.

Five dose levels will be examined, starting at the lowest, in each population with 10 participants in each dose level. These participants will be randomized to receive TAK-063 (8 subjects) and placebo (2 subjects) once daily (QD) for 7 days.

In total, approximately 60 participants will be enrolled in the study. This trial will be conducted in single site in the United States. The overall time to participate in this study is up to 42 days. Participants will make 2 visits to the clinic, including 8-10 days confinement to the clinic, and will be contacted by telephone 7 days after last dose of study drug for a follow-up assessment.

Dose escalation and the actual choice of the subsequent dose level will only occur following a review of the blinded data from the previous cohorts.

ELIGIBILITY:
Inclusion Criteria:

Healthy Participants:

1. Aged 20-55 years, inclusive, at the time of informed consent and first study medication dose.
2. Is a healthy adult male or female of Japanese descent (born to Japanese parents and grandparents and has lived outside of Japan for less than 5 years).
3. Weighs at least 45 kg and has a body mass index (BMI) between 18.0 and 28.0 kg/m^2, inclusive, at Screening.

Participants with Stable Schizophrenia:

1. Is aged 18 to 55 years, inclusive, at the time of informed consent and first study medication dose.
2. Is an adult male or female with a diagnosis of schizophrenia or schizoaffective disorder.
3. Weighs at least 45 kg and has a BMI between 18.0 and 35.0 kg/m^2, inclusive at Screening.
4. Has been receiving a stable dose of antipsychotic monotherapy for at least 1 month prior to Screening.
5. Has not had an acute exacerbation of psychosis or been hospitalization for the treatment of schizophrenia or schizoaffective disorder for at least 3 months prior to Screening.

Exclusion Criteria:

All Participants:

1. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality (other than the disease being studied), which may impact the ability of the participant to participate or potentially confound the study results.
2. If female, the participant is pregnant or lactating or intending to become pregnant, or intending to donate ova, before, during the course of the study or within 12 weeks after last dose.
3. Intends to donate sperm during the course of this study or for 12 weeks after last dose.
4. Has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking TAK-063, or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.

Healthy Participants:

1. Has a history or treatment of Axis I/II mental disorders according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) such as depression, anxiety disorders, bipolar disorder, attention deficit hyperactivity disorder (ADHD), autism spectrum disorders, anorexia nervosa, bulimia nervosa or schizophrenia within the past 3 years.
2. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in Day -1. Cotinine test is positive at Screening or Check-in (Day -1).

Participants with Stable Schizophrenia:

1. Has a history of a primary DSM-IV axis I diagnosis other than schizophrenia or schizoaffective disorder.
2. Has not discontinued antipsychotic or other psychotropic medications or is unable to discontinue antipsychotic or other psychotropic medications at Day -7 (or five half-lives prior to Day -1).
3. Is taking a concomitant medication for a medical condition at a stable dose or regimen for less than two months or is taking a concomitant medication for a medical condition for less than two months and for which the discontinuation for the study period is not medically permissible.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Glendale, California, United States

REFERENCES:
- [Derived] Goldsmith P, Affinito J, McCue M, Tsai M, Roepcke S, Xie J, Gertsik L, Macek TA. A Randomized Multiple Dose Pharmacokinetic Study of a Novel PDE10A Inhibitor TAK-063 in Subjects with Stable Schizophrenia and Japanese Subjects and Modeling of Exposure Relationships to Adverse Events. Drugs R D. 2017 Dec;17(4):631-643. doi: 10.1007/s40268-017-0214-8. PMID 29103081

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 21 June 2013 (First participant signed consent) to 23 June 2014.
Pre-assignment Details: Participants with a diagnosis of Schizophrenia were enrolled into 1 of 6 treatment groups, once a day placebo, 3 mg, 10 mg, 20 mg, 30 mg or 100 mg TAK-063. Healthy Japanese participants were enrolled in 1 of 4 treatment groups, once a day placebo, 3 mg, 10 mg or 20 mg TAK-063.
Groups:
- TAK-063 3 mg (Schizophrenia Participants): TAK-063 3 mg, tablets, orally, once daily for 7 days in participants with Schizophrenia.
- TAK-063 10 mg (Schizophrenia Participants): TAK-063 10 mg, tablets, orally, once daily for 7 days in participants with Schizophrenia.
- TAK-063 20 mg (Schizophrenia Participants): TAK-063 20 mg, tablets, orally, once daily for 7 days in participants with Schizophrenia.
- TAK-063 30 mg (Schizophrenia Participants): TAK-063 30 mg, tablets, orally, once daily for 7 days in participants with Schizophrenia.
- TAK-063 100 mg (Schizophrenia Participants): TAK-063 100 mg, tablets, orally, once daily for 7 days in participants with Schizophrenia.
- Placebo (Schizophrenia Participants): Placebo matching TAK-063, tablets, orally, once daily for 7 days in participants with Schizophrenia.
- TAK-063 3 mg (Healthy Participants): TAK-063 3 mg, tablets, orally, once daily for 7 days in healthy Japanese participants.
- TAK-063 10 mg (Healthy Participants): TAK-063 10 mg, tablets, orally, once daily for 7 days in healthy Japanese participants.
- TAK-063 20 mg (Healthy Participants): TAK-063 20 mg, tablets, orally, once daily for 7 days in healthy Japanese participants.
- Placebo (Healthy Participants): Placebo matching TAK-063, tablets, orally, once daily for 7 days in healthy Japanese participants.
Period: Overall Study
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | Placebo (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants) | Placebo (Healthy Participants)
Started | 7 | 8 | 7 | 8 | 8 | 9 | 8 | 8 | 8 | 6
Completed | 7 | 7 | 7 | 7 | 7 | 9 | 8 | 7 | 6 | 6
Not Completed | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0
Not completed — Pretreatment Event/Adverse Event | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Voluntary Withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | Placebo (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants) | Placebo (Healthy Participants) | Total
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 8 | 9 | 8 | 8 | 8 | 6 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (4.20) | 39.6 (9.90) | 44.6 (9.00) | 45.3 (8.19) | 39.4 (8.14) | 43.1 (11.34) | 36.3 (9.78) | 25.9 (9.51) | 34.6 (10.61) | 38.5 (11.52) | 39.0 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 (NA) | 4 (NA) | 1 (NA) | 3 (NA) | 1 (NA) | 4 | 2 (9.78) | 0 (9.51) | 0 (10.61) | 1 (11.52) | 19
  Male | 4 | 4 | 6 | 5 | 7 | 5 | 6 | 8 | 8 | 5 | 58
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4
  Non-Hispanic or Latino | 6 | 7 | 7 | 8 | 7 | 8 | 8 | 8 | 8 | 6 | 73
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 8 | 8 | 8 | 6 | 31
  Black or African American | 6 | 5 | 4 | 7 | 7 | 8 | 0 | 0 | 0 | 0 | 37
  White | 1 | 3 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 8
  Multiracial | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 7 | 8 | 8 | 9 | 8 | 8 | 8 | 6 | 77
Height [Mean (Standard Deviation); unit: cm] | 172.1 (9.19) | 166.8 (7.89) | 172.6 (9.61) | 166.3 (7.70) | 173.9 (8.82) | 173.3 (10.95) | 172.5 (10.35) | 170.5 (7.21) | 171.8 (7.46) | 168.8 (6.49) | 171.0 (8.44)
Weight [Mean (Standard Deviation); unit: kg] | 92.09 (10.138) | 74.75 (8.543) | 83.76 (19.701) | 88.83 (12.805) | 83.51 (11.853) | 86.46 (17.422) | 73.98 (10.503) | 67.45 (8.128) | 70.19 (6.879) | 63.50 (10.037) | 78.70 (14.666)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.13 (3.266) | 26.98 (3.476) | 27.93 (5.488) | 32.16 (4.243) | 27.76 (4.460) | 28.80 (5.710) | 24.75 (1.962) | 22.65 (2.556) | 24.14 (1.984) | 22.23 (2.778) | 26.93 (4.812)
Caffeine Consumption [Number; unit: participants]
  Yes | 3 | 8 | 5 | 5 | 2 | 8 | 3 | 4 | 6 | 3 | 47
  No | 4 | 0 | 2 | 3 | 6 | 1 | 5 | 4 | 2 | 3 | 30
Smoking Classification [Number; unit: participants]
  Never smoked | 0 | 1 | 0 | 2 | 0 | 1 | 7 | 2 | 5 | 2 | 20
  Current smoker | 5 | 7 | 6 | 5 | 7 | 8 | 0 | 0 | 0 | 0 | 38
  Ex-smoker | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 6 | 3 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience at Least One Treatment-Emergent Adverse Event (TEAE) After 7 Days of Dosing
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Day 1 to Day 14
Population: Safety population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | Placebo (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants) | Placebo (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 8 | 9 | 8 | 8 | 8 | 6
percentage of participants | 57.1 | 87.5 | 71.4 | 75.0 | 100.0 | 55.6 | 50.0 | 62.5 | 62.5 | 50.0

2. Primary Outcome: Percentage of Participants With Markedly Abnormal Safety Laboratory Tests
Description: The percentage of participants with any markedly abnormal standard safety laboratory values, including hematology, serum chemistries, and urinalysis, during the treatment period.
Time Frame: Day 1 to Day 8
Population: Safety population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | Placebo (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants) | Placebo (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 8 | 9 | 8 | 8 | 8 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 25.0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Markedly Abnormal Vital Sign Measurements
Description: The percentage of participants who meet markedly abnormal criteria for vital signs, including oral body temperature, respiration rate, pulse, and resting blood pressure and after standing
Time Frame: Day 1 to Day 8
Population: Safety population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | Placebo (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants) | Placebo (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 8 | 9 | 8 | 8 | 8 | 6
percentage of participants | 71.4 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

4. Primary Outcome: Percentage of Participants With Markedly Abnormal Values of 12-Lead Electrocardiogram (ECG) Parameters
Description: The percentage of participants who meet markedly abnormal criteria specified by the protocol and statistical analysis plan during the treatment period.
Time Frame: Day 1 to Day 8
Population: Safety population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | Placebo (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants) | Placebo (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 8 | 9 | 8 | 8 | 8 | 6
percentage of participants | 57.1 | 50.0 | 57.1 | 75.0 | 62.5 | 44.4 | 50.0 | 75.0 | 50.0 | 33.3

5. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-063 and TAK-063 Metabolite M-I
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Days 1 and 7 pre-dose and multiple time-points post-dose (Up to 24 hours)
Population: PK Set included all randomized participants who received study drug for whom PK data was available for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 8
ng/mL
  TAK-063 Day 1 | 17.0 (7.2) | 62.8 (16.6) | 95.1 (30.8) | 151.4 (31.9) | 211.3 (84.8) | 14.9 (5.3) | 69.4 (13.2) | 116.2 (17.9)
  TAK-063 M-I Day 1 | 11.3 (4.2) | 64.8 (21.5) | 98.5 (29.1) | 93.2 (4.8) | 126.7 (29.9) | 8.8 (1.7) | 36.0 (5.0) | 61.8 (11.2)
  TAK-063 Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 25.6 (4.6) | 70.3 (11.5) | 120.0 (39.3) | 179.4 (34.9) | 228.3 (55.1) | 29.1 (8.0) | 74.6 (12.5) | 139.8 (25.4)
  TAK-063 M-I Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 19.2 (4.2) | 74.8 (20.3) | 123.6 (48.2) | 108.5 (15.8) | 127.7 (22.6) | 15.1 (2.4) | 38.2 (4.4) | 70.9 (17.8)

6. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-063 and TAK-063 Metabolite M-I
Description: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: Days 1 and 7 pre-dose and multiple time-points post-dose (Up to 24 hours)
Population: PK Set included all randomized participants who received study drug for whom PK data was available for analysis.
Measure: Median (Full Range); unit: hour
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 8
hour
  TAK-063 Day 1 | 3.0 [1.0 to 6.0] | 2.0 [1.5 to 4.0] | 3.0 [3.0 to 3.0] | 3.0 [2.0 to 4.0] | 4.0 [2.0 to 6.0] | 3.0 [1.5 to 4.0] | 3.0 [2.0 to 8.0] | 2.5 [1.5 to 4.0]
  TAK-063 M-I Day 1 | 3.0 [1.0 to 6.0] | 2.0 [1.5 to 6.0] | 3.0 [3.0 to 4.0] | 3.1 [2.0 to 6.5] | 3.0 [2.0 to 6.0] | 2.5 [1.5 to 4.0] | 3.0 [2.0 to 6.0] | 3.0 [1.5 to 4.0]
  TAK-063 Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 3.0 [2.0 to 6.0] | 3.0 [1.0 to 6.0] | 3.0 [2.0 to 4.0] | 3.0 [1.5 to 3.0] | 3.0 [2.0 to 3.3] | 3.0 [1.5 to 4.0] | 1.5 [1.0 to 6.0] | 2.5 [1.5 to 4.0]
  TAK-063 M-I Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 4.0 [2.0 to 6.0] | 3.0 [1.5 to 6.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [1.5 to 6.0] | 3.0 [3.0 to 4.0]

7. Secondary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-063 and TAK-063 Metabolite M-I
Description: AUC(0-tlqc) is a measure of total plasma exposure to the drug from time 0 to time of the Last Quantifiable Concentration.
Time Frame: Days 1 and 7 pre-dose and multiple time-points post-dose (Up to 24 hours)
Population: PK Set included all randomized participants who received study drug for whom PK data was available for analysis.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 8
ng*hr/mL
  TAK-063 Day 1 | 158.8 (59.8) | 622.7 (140.9) | 938.3 (401.0) | 1616.6 (392.1) | 2499.3 (1143.3) | 148.3 (54.8) | 651.3 (73.2) | 1242.3 (275.4)
  TAK-063 M-I Day 1 | 113.9 (48.9) | 681.8 (268.9) | 1009.6 (516.5) | 1069.1 (120.2) | 1481.1 (404.5) | 74.7 (19.1) | 327.6 (37.4) | 666.3 (148.8)
  TAK-063 Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 280.8 (60.4) | 680.3 (153.4) | 1240.9 (385.4) | 2030.9 (479.2) | 2764.5 (711.4) | 295.6 (83.5) | 736.1 (90.7) | 1536.7 (236.7)
  TAK-063 M-I Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 218.9 (56.9) | 786.3 (296.6) | 1387.2 (681.0) | 1371.2 (291.8) | 1598.8 (288.7) | 156.7 (37.3) | 378.5 (51.6) | 806.5 (174.3)

8. Secondary Outcome: AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Postdose for TAK-063 and TAK-063 Metabolite M-I
Description: AUC(0-24) is a measure of total plasma exposure to the drug from Time 0 to 24 hours post-dose.
Time Frame: Days 1 and 7 pre-dose and multiple time-points post-dose (Up to 24 hours)
Population: PK Set included all randomized participants who received study drug for whom PK data was available for analysis.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 8
ng*hr/mL
  TAK-063 Day 1 | 159.0 (60.0) | 623.2 (141.0) | 939.3 (402.0) | 1619.0 (393.3) | 2503.2 (1146.4) | 148.6 (54.9) | 651.9 (73.3) | 1243.9 (276.0)
  TAK-063 M-I Day 1 | 114.0 (49.1) | 682.5 (269.0) | 1011.0 (517.9) | 1070.8 (120.7) | 1483.6 (405.8) | 74.8 (19.2) | 327.9 (37.5) | 667.3 (149.1)
  TAK-063 Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 280.6 (60.5) | 680.1 (153.3) | 1240.9 (385.4) | 2030.9 (479.2) | 2764.0 (712.1) | 295.6 (83.5) | 736.1 (90.6) | 1536.4 (236.2)
  TAK-063 M-I Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 218.7 (57.0) | 786.0 (296.4) | 1387.2 (681.0) | 1371.2 (291.8) | 1598.4 (289.1) | 156.7 (37.3) | 378.5 (51.6) | 806.3 (174.1)

9. Secondary Outcome: CL/F: Oral Clearance of TAK-063
Description: CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided by area under the curve from time 0 to 24 hours post-dose, after multiple dosing (at steady state).
Time Frame: Days 1 and 7 pre-dose and multiple time-points post-dose (Up to 24 hours)
Population: PK Set included all randomized participants who received study drug for whom PK data was available for analysis.
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 8
liter/hour
  TAK-063 Day 1 | 16.1 (7.3) | 14.0 (4.3) | 21.3 (8.0) | 14.4 (5.4) | 38.1 (25.0) | 16.9 (5.2) | 13.9 (2.0) | 13.9 (4.6)
  TAK-063 Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 11.2 (2.7) | 15.4 (3.9) | 17.1 (4.0) | 15.5 (3.5) | 38.5 (10.8) | 10.8 (2.8) | 13.8 (1.6) | 13.3 (1.9)

10. Secondary Outcome: Average Plasma Concentration on Day 1 (Cav) and Day 7 (Cavss) for TAK-063 and TAK-063 Metabolite M-I
Description: Cav is the Average plasma concentration on Day 1, calculated as AUC(0-24)/24 on Day 1. Cavss is the average plasma concentration on Day 7, calculated as AUC(0-24)/24 on Day 7.
Time Frame: Days 1 and 7 pre-dose and multiple time-points post-dose (Up to 24 hours)
Population: PK Set included all randomized participants for whom PK data was available for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 8
ng/mL
  TAK-063 Day 1 | 6.6 (2.5) | 26.0 (5.9) | 39.1 (16.8) | 67.5 (16.4) | 104.3 (47.8) | 6.2 (2.3) | 27.2 (3.1) | 51.8 (11.5)
  TAK-063 M-I Day 1 | 4.8 (2.0) | 28.4 (11.2) | 42.1 (21.6) | 44.6 (5.0) | 61.8 (16.9) | 3.1 (0.8) | 13.7 (1.6) | 27.8 (6.2)
  TAK-063 Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 11.7 (2.5) | 28.3 (6.4) | 51.7 (16.1) | 84.6 (20.0) | 115.2 (29.7) | 12.3 (3.5) | 30.7 (3.8) | 64.0 (9.8)
  TAK-063 M-I Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 9.1 (2.4) | 32.8 (12.4) | 57.8 (28.4) | 57.1 (12.2) | 66.6 (12.0) | 6.5 (1.6) | 15.8 (2.2) | 33.6 (7.3)

11. Secondary Outcome: Cmax Molar Ratio: Ratio of TAK-063 Metabolite Cmax to TAK-063 Cmax
Description: Cmax Molar Ratio is the ratio of Cmax molar values of the metabolite compared to the parent calculated by dividing Cmax molar values of metabolite M-I with those of TAK-063.
Time Frame: Days 1 and 7 pre-dose and multiple time-points post-dose (Up to 24 hours)
Population: PK Set included all randomized participants who received study drug for whom PK data was available for analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 8
ratio
  TAK-063 M-I Day 1 | 0.7 (0.1) | 1.0 (0.2) | 1.0 (0.2) | 0.6 (0.1) | 0.6 (0.2) | 0.6 (0.2) | 0.5 (0.1) | 0.5 (0.1)
  TAK-063 M-I Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 0.7 (0.2) | 1.0 (0.2) | 1.0 (0.2) | 0.6 (0.1) | 0.6 (0.1) | 0.5 (0.1) | 0.5 (0.1) | 0.5 (0.1)

12. Secondary Outcome: AUC(0-24) Ratio: Ratio of TAK-063 Metabolite AUC(0-24) to TAK-063 AUC(0-24)
Description: AUC(0-24) Ratio is the ratio of AUC(0-24) values of the metabolite compared to the parent calculated by dividing AUC(0-24) values of metabolite M-I with those of the parent drug TAK-063.
Time Frame: Days 1 and 7 pre-dose and multiple time-points post-dose (Up to 24 hours)
Population: PK Set included all randomized participants who received study drug for whom PK data was available for analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 8
ratio
  TAK-063 M-I Day 1 | 0.7 (0.1) | 1.0 (0.3) | 1.0 (0.2) | 0.7 (0.1) | 0.6 (0.2) | 0.5 (0.1) | 0.5 (0.1) | 0.5 (0.1)
  TAK-063 M-I Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 0.8 (0.2) | 1.1 (0.3) | 1.1 (0.2) | 0.7 (0.1) | 0.6 (0.1) | 0.5 (0.04) | 0.5 (0.1) | 0.5 (0.1)

13. Secondary Outcome: Accumulation Ratios Between Day 7 AUC(0-24) and Day 1 AUC(0-24)
Description: Accumulation ratios between Day 7 AUC(0-24) and Day 1 AUC(0-24), (Day 7/Day 1). Estimated Ratio (Day 7/Day 1) is the exponentiated results of the difference between Day 7 and Day 1 in log-transformed values which resolves to the ratio of Day 7/Day 1 estimates.
Time Frame: Days 1 and 7 pre-dose and multiple time-points post-dose (Up to 24 hours)
Population: PK Set included all randomized participants who received study drug for whom PK data was available for analysis.
Measure: Mean (90% Confidence Interval); unit: ratio
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants)
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 8 | 7 | 6
ratio
  TAK-063 | 1.8 (0.550) [1.6 to 2.1] | 1.1 (0.210) [1.0 to 1.3] | 1.4 (0.325) [1.2 to 1.6] | 1.3 (0.126) [1.1 to 1.5] | 1.2 (0.324) [1.0 to 1.4] | 2.0 (0.472) [1.8 to 2.3] | 1.1 (0.169) [1.0 to 1.3] | 1.2 (0.180) [1.0 to 1.3]
  TAK-063 M-I | 2.0 (0.619) [1.7 to 2.4] | 1.2 (0.308) [1.0 to 1.4] | 1.4 (0.371) [1.2 to 1.6] | 1.3 (0.183) [1.1 to 1.5] | 1.1 (0.243) [0.9 to 1.3] | 2.1 (0.408) [1.9 to 2.3] | 1.1 (0.158) [1.0 to 1.3] | 1.1 (0.226) [1.0 to 1.3]

14. Secondary Outcome: Ae(0-24): Total Amount Excreted in the Urine From Time 0 to 24 Hours Postdose for TAK-063 and TAK-063 Metabolite M-I
Description: Ae(0-24) is a measure of the total amount of study drug excreted in the urine from time 0 to 24 hours postdose.
Time Frame: Days 1 and 7 pre-dose and multiple time-points post-dose (Up to 24 hours)
Population: PK Set included all randomized participants who received study drug for whom PK data was available for analysis.
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 8
ng
  TAK-063 Day 1 | 0.0 (0.0) | 3642.3 (2611.9) | 4432.8 (3418.6) | 9952.1 (6025.2) | 34893.4 (27402.5) | 0.0 (0.0) | 3592.0 (4936.1) | 14145.4 (9576.1)
  TAK-063 M-I Day 1 | 0.0 (0.0) | 9099.4 (3451.0) | 16879.5 (8061.5) | 24302.0 (12756.6) | 52682.9 (14870.1) | 0.0 (0.0) | 10487.8 (5847.3) | 26557.0 (11839.7)
  TAK-063 Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 0.0 (0.0) | 4430.9 (2831.5) | 7979.2 (4739.0) | 15066.0 (9996.7) | 35527.5 (20919.1) | 0.0 (0.0) | 4765.2 (3491.0) | 15913.7 (9619.6)
  TAK-063 M-I Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 630.2 (1129.4) | 11708.6 (7047.1) | 25327.7 (12723.6) | 35462.0 (11737.9) | 67767.6 (36686.1) | 1024.2 (1665.5) | 14139.9 (8205.9) | 35341.3 (12664.4)

15. Secondary Outcome: Fe: Fraction of Drug Excreted in Urine for TAK-063
Description: Fe is a measure of the fraction of drug excreted in urine and is calculated as Fe = (total amount excreted in the urine from time 0 to 24 hours post-dose / dose)×100
Time Frame: Days 1 and 7 pre-dose and multiple time-points post-dose (Up to 24 hours)
Population: PK Set included all randomized participants who received study drug for whom PK data was available for analysis.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants)
Number analyzed (Participants) | 7 | 8 | 7 | 8 | 7 | 8 | 8 | 8
percent
  Day 1 | 0.00 (0.00) | 0.04 (0.03) | 0.02 (0.02) | 0.03 (0.02) | 0.03 (0.03) | 0.00 (0.00) | 0.04 (0.05) | 0.07 (0.05)
  Day 7 (n=7, 7, 7, 7, 7, 8, 7, 6) | 0.00 (0.00) | 0.04 (0.03) | 0.04 (0.02) | 0.05 (0.03) | 0.04 (0.02) | 0.00 (0.00) | 0.05 (0.03) | 0.08 (0.05)

16. Secondary Outcome: CLr: Renal Clearance of TAK-063 and TAK-063 Metabolite M-I
Description: CLr is a measure of apparent clearance of the drug from the urine calculated as total amount excreted in the urine from time 0 to 24 hours postdose / plasma area under the curve from time 0 to 24 hours post-dose.
Time Frame: Days 1 and 7 pre-dose and multiple time-points post-dose (Up to 24 hours)
Population: PK Set included all randomized participants who received study drug for whom PK data was available for analysis.
Measure: Mean (Standard Deviation); unit: mL/hour
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants)
Number analyzed (Participants) | 2 | 8 | 6 | 7 | 7 | 3 | 7 | 8
mL/hour
  TAK-063 Day 1 (n=0, 6, 6, 7, 7, 0, 6, 7) | NA (NA) — CLr could not be calculated because the concentrations in urine were low/not detected. | 8.4 (3.9) | 5.2 (2.5) | 6.7 (1.6) | 16.2 (13.1) | NA (NA) — CLr could not be calculated because the concentrations in urine were low/not detected. | 7.0 (7.0) | 12.9 (7.5)
  TAK-063 M-I Day 1 (n=0, 8, 6, 7, 7, 0, 7, 8) | NA (NA) — CLr could not be calculated because the concentrations in urine were low/not detected. | 15.9 (10.7) | 20.4 (8.0) | 25.6 (9.3) | 36.8 (11.9) | NA (NA) — CLr could not be calculated because the concentrations in urine were low/not detected. | 38.0 (16.4) | 39.9 (16.1)
  TAK-063 Day 7 (n=0, 7, 6, 7, 7, 0, 6, 6) | NA (NA) — CLr could not be calculated because the concentrations in urine were low/not detected. | 6.8 (4.4) | 7.2 (1.1) | 7.3 (3.4) | 13.3 (7.3) | NA (NA) — CLr could not be calculated because the concentrations in urine were low/not detected. | 7.3 (3.2) | 10.5 (6.3)
  TAK-063 M-I Day 7 (n=2, 7, 6, 7, 7, 3, 6, 6) | 11.3 (6.7) | 16.9 (15.5) | 21.7 (8.8) | 26.4 (8.7) | 41.4 (17.0) | 14.2 (6.8) | 42.8 (14.0) | 45.5 (17.5)

ADVERSE EVENTS:
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-063 3 mg (Schizophrenia Participants) | TAK-063 10 mg (Schizophrenia Participants) | TAK-063 20 mg (Schizophrenia Participants) | TAK-063 30 mg (Schizophrenia Participants) | TAK-063 100 mg (Schizophrenia Participants) | Placebo (Schizophrenia Participants) | TAK-063 3 mg (Healthy Participants) | TAK-063 10 mg (Healthy Participants) | TAK-063 20 mg (Healthy Participants) | Placebo (Healthy Participants)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/7 | 0/8 | 0/8 | 0/9 | 0/8 | 0/8 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 4/7 | 7/8 | 5/7 | 6/8 | 8/8 | 5/9 | 4/8 | 5/8 | 5/8 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-063 3 mg (Schizophrenia Participants) (N=7) | TAK-063 10 mg (Schizophrenia Participants) (N=8) | TAK-063 20 mg (Schizophrenia Participants) (N=7) | TAK-063 30 mg (Schizophrenia Participants) (N=8) | TAK-063 100 mg (Schizophrenia Participants) (N=8) | Placebo (Schizophrenia Participants) (N=9) | TAK-063 3 mg (Healthy Participants) (N=8) | TAK-063 10 mg (Healthy Participants) (N=8) | TAK-063 20 mg (Healthy Participants) (N=8) | Placebo (Healthy Participants) (N=6)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Catheter Site Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling Of Body Temperature Change (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic Heart Rate Response Increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 3 | 4 | 4 | 8 | 2 | 3 | 4 | 5 | 2
Akathisia (Nervous system disorders) | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Extrapyramidal Disorder (Nervous system disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0
Oromandibular Dystonia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dizziness Postural (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dystonia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disturbance In Attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menopausal Symptoms (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vessel Puncture Site Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nail Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.